CLINICAL TRIAL: NCT03320460
Title: Efficacy of Photobiomodulation for Oral Lichen Planus Treatment
Brief Title: Photobiomodulation in Oral Lichen Planus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Maria Fernanda Setúbal Destro Rodrigues, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.375.410
Record Dates: First submitted 2017-10-17; First posted 2017-10-25 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Lichen Planus, Oral; Low-Level Light Therapy
Keywords: oral lichen planus; photobiomodulation; inflammation
MeSH Terms: conditions — Lichen Planus, Oral; Inflammation | interventions — Clobetasol; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Control group Experimental Group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Control group will be treated with clobetasol propionate 0.05% gel for 30 consecutive days and the laser device will be positioned over the lesion but will be switched off to mask the treatment. The experimental group will be treated with placebo gel for 30 consecutive days to mask the treatment and patients will receive laser treatment twice a week during 1 month for PBM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental): Patients will be treated with localized PBM with a diode laser with continuous wave (laser λ =660 nm; power 100mW;radiant energy: 177J/cm2; 5-s exposure time per point and 0.5J of energy per point) applied directly to the surrounding oral mucosa and to the center of OLP, always by the same operator, twice a week for 4 weeks, totaling 8 session. The number of points will be variable according to the lesion size. The output power of the laser equipment will be evaluated using a power meter (Laser Check; MMOptics LTDA, São Paulo, Brazil) before treatment to confirm the effective mean power as well as the doses applied during the procedure.
  Interventions: Device: Photobiomodulation; Other: Placebo gel
- Propionate clobetasol gel 0.05% (Active Comparator): Patients will be treated with Propionate clobetasol gel 0.05% for 30 consecutive days. Laser device will be positioned over the lesion but will be switched off to mask the treatment. Patients will be instructed to apply the propionate clobetasol gel 0.05% in the entire lesion three times/days. To prevent oral candidiasis, patients will use micostatin solution (Nystatin oral suspension 100,000 USP/ml) once a day during 4 weeks.
  Interventions: Drug: Propionate clobetasol gel 0.05%; Other: Placebo Photobiomodulation

INTERVENTIONS:
Drug: Propionate clobetasol gel 0.05% — Patients will be treated with Propionate clobetasol gel 0.05% for 30 consecutive days and with placebo laser twice a week. Patients will be instructed to apply the propionate clobetasol gel 0.05% in the entire lesion three times/days. To prevent oral candidiasis, patients will use micostatin solution (Nystatin oral suspension 100,000 USP/ml) once a day during 4 weeks.
  Other Names: Clobetasol
  Arms: Propionate clobetasol gel 0.05%
Device: Photobiomodulation — Patients will be treated with localized PBM with a diode laser with continuous wave (laser λ = 660 nm; power 100mW;radiant energy: 177J/cm2; 5-s exposure time per point and 0.5J of energy per point) applied directly to the surrounding oral mucosa and to the center of OLP, always by the same operator, twice a week for 4 weeks, totaling 8 session. The number of points will be variable according to the lesion size. The output power of the laser equipment will be evaluated using a power meter (Laser Check; MMOptics LTDA, São Paulo, Brazil) before treatment to confirm the effective mean power as well as the doses applied during the procedure.
  Other Names: Low level laser therapy
  Arms: Photobiomodulation
Other: Placebo gel — Placebo gel for 30 consecutive days to mask the treatment
  Other Names: inative gel
  Arms: Photobiomodulation
Other: Placebo Photobiomodulation — Laser device will be positioned over the lesion but will be switched off to mask the treatment.
  Other Names: Laser off
  Arms: Propionate clobetasol gel 0.05%

SUMMARY:
The aim of this study was to compare the efficacy of PBM (660nm) and corticosteroid therapy with clobetasol propionate 0.05% in the treatment of OLP. This is a protocol for a randomized, controlled, double blind clinical trial. Fourty-four patients will be randomized in two experimental groups. Control group will be treated with clobetasol propionate 0.05% for 30 consecutive days and with placebo PBM twice a week. The experimental group will be treated with placebo gel for 30 consecutive days to mask the treatment and patients will receive PBM twice a week during 1 month (laser λ = 660±10 nm; power 100mW; radiant energy 177J/cm2; 5-s exposure time per point and 0.5J of energy per point. The primary variable (pain) and the secondary variables including clinical scores and functional scores as well as patient anxiety and depression (The Hospital Anxiety and Depression Scale-HADS), will be evaluated at the baseline, once a week during treatment and after 30 and 60 days of follow up. Evaluation of clinical resolution will be performed at the end of the treatment (30 days). Evaluation of recurrence will be performed after 30 and 60 days of follow up. Serum and salivary levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated at baseline and at the end of treatment (30 days). Quality of life will be evaluated by OHIP-14 questionnaire at baseline, at the end of treatment and after 30 and 60 days of follow up. The chi-square test, Student's t-test and ANOVA will be used and the level of significance of 5% will be considered (p < 0.05).

DETAILED DESCRIPTION:
Oral lichen planus is an idiopathic chronic mucocutaneous disease with a ride range of clinical manifestations, including white reticular patches, erosive/ulcerative and atrophic lesions, both associated with intense symptomatology. CD4+ and CD8+ T lymphocytes cells play an important role in the pathogenesis of OLP and are responsible for the production of different cytokines, including IL-6, IL-10, IL-1β, INF-γ and TNF-α. Treatment is symptomatic and topical corticosteroids are commonly used as standard therapy. However, patients frequently present relapses after treatment's discontinuation, develop resistance to corticosteroids therapy as well as secondary candidiasis. Photobiomodulation (PBM) has shown to be a potential therapeutic tool to treat inflammatory disorders, including OLP. Some studies have demonstrated that PBM improves the clinical presentation of OLP (erosive/ulcerative or atrophic lesions to reticular lesions), reduces pain and recurrence. However, it remains controversy if PBM is more effective than corticosteroid in the treatment of OLP. The aim of this study is to evaluate the efficacy of PBM in the treatment of OLP in relation to the standard therapy with corticosteroids. This is a protocol for a randomized, controlled, doubled blind clinical trial, with two months of follow up.

Patients with symptomatic OLP and with histopathological diagnosis of OLP based on WHO criteria will be included in this study. Fourty-four patients will be randomized in two experimental groups. Control group will be treated with clobetasol propionate 0.05% gel for 30 consecutive days and the laser device will be positioned over the lesion but will be switched off to mask the treatment. The experimental group will be treated with placebo gel for 30 consecutive days to mask the treatment and patients will receive laser treatment twice a week during 1 month for PBM (laser λ = 660±10 nm; power 100mW; radiant energy; 177J/cm2; 5-s exposure time per point and 0.5J of energy per point). The primary variable (pain by VAS scale) and the secondary variables (clinical scores, functional scores and Patient anxiety and depression) will be evaluated at the baseline, once a week during treatment and after 30 and 60 days of follow up. Evaluation of clinical resolution will be performed at the end of the treatment (30 days). Evaluation of recurrence will be performed after 30 and 60 days of follow up. Serum and salivary levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated at baseline and at the end of treatment (30 days). Quality of life will be evaluated by OHIP-14 questionnaire at baseline, at the end of treatment and after 30 and 60 days of follow up. The findings will be computed and submitted to statistical analysis. Interval estimates will be used for the variables of interest to determine the prevision of the estimates and perform comparisons. If necessary, transformation methods or non-parametric tests will be applied. The chi-square test, Student's t-test and ANOVA will be used and the level of significance of 5% will be considered (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* The participants in this study will be male and female (aged over 18 years) diagnosed with symptomatic oral lichen planus, based on the clinical and histopathological criteria of the World Health Organization (WHO).

Exclusion Criteria:

* Patients with ongoing cancer; pregnant or breastfeeding women; patients with history of corticosteroids and nonsteroidal anti-inflammatory treatment in the last one months, patients with uncontrolled systemic disease; consumption of illicit drugs; use of medication associated with oral lichenoid reactions; amalgam restoration near to OLP lesions; epithelial dysplasia in the histopathological examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain of OLP | Participants will be evaluated at baseline (Day 0)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | Participants will be evaluated after 1 week of treatment (Day 7)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | Participants will be evaluated after 2 weeks of treatment (Day 14)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | Participants will be evaluated after 3 weeks of treatment (Day 21)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | Participants will be evaluated after 4 weeks of treatment (Day 30)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | 30 days after the discontinuation of treatment (follow-up period)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Assessment of Pain of OLP | 60 days after the discontinuation of treatment (follow-up period)
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.

SECONDARY OUTCOMES:
Assessment of clinical presentation of OLP | Participants will be evaluated at baseline (Day 0)
  Clinical data will be evaluated by scores according to Thongprasom et al
Assessment of clinical presentation of OLP | Participants will be evaluated after 1 week of treatment (Day 7)
  Clinical data will be evaluated by scores according to Thongprasom et al
Assessment of clinical presentation of OLP | Participants will be evaluated after 2 weeks of treatment (Day 14)
  Clinical data will be evaluated by scores according to Thongprasom et al
Assessment of clinical presentation of OLP | Participants will be evaluated after 3 weeks of treatment (Day 21)
  Clinical data will be evaluated scores according to Thongprasom et al
Assessment of clinical presentation of OLP | Participants will be evaluated after 4 weeks of treatment (Day 30)
  Clinical data will be evaluated by scores according to Thongprasom et al
Assessment of clinical presentation of OLP | 30 days after the discontinuation of treatment (follow-up period)
  Clinical data will be evaluated by scores according to Thongprasom et al
Assessment of clinical presentation of OLP | 60 days after the discontinuation of treatment (follow-up period)
  Clinical data will be evaluated by scores according to Thongprasom et al
Function | Participants will be evaluated at baseline (Day 0)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | Participants will be evaluated after 1 week of treatment (Day 7)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | Participants will be evaluated after 2 weeks of treatment (Day 14)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | Participants will be evaluated after 3 weeks of treatment (Day 21)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | Participants will be evaluated after 4 weeks of treatment (Day 30)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | 30 days after the discontinuation of treatment (follow-up period)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Function | 60 days after the discontinuation of treatment (follow-up period)
  The functional scores will be applied to evaluate chewing function, swallowing, fluid intake and altered sense of taste, according to Libelly et al (2006). Each function evaluated will receive the follow scores: 0 ( no difficulty) , 1 ( mild difficulty) , 2, ( moderate difficulty), 3, (severe difficulty), and 4 ( impossibility to perform certain function).
Clinical Resolution | Participants will be evaluated after 4 weeks of treatment (Day 30)
  The clinical resolution will be evaluated at the end of treatment (day 30) according to Corozzo et al. (1999). Complete resolution will be considered when patients present absence of symptoms and remission of atrophic/erosive lesions regardless the presence of any persisting hyperkeratotic lesions. Partial resolution will be considered when a decrease but not the complete remission of atrophic/erosive areas and symptoms were observed. No response to treatment will be considered when OLP lesions present the same clinical or worse presentation in relation to the baseline condition.
Recurrence rate | The recurrence rate will be evaluated 30 days after the discontinuation of treatment (follow-up period)
  No recurrence will be considered when the patient presents the same clinical aspect of lesion at the end of treatment and recurrence, when the patient present new atrophic/erosive lesion at the same site during the follow-up period.
Recurrence rate | The recurrence rate will be evaluated 60 days after the discontinuation of treatment (follow-up period)
  No recurrence will be considered when the patient presents the same clinical aspect of lesion at the end of treatment and recurrence, when the patient present new atrophic/erosive lesion at the same site during the follow-up period.
Salivary levels of IL-1β, IL-6, IL-8, IL-10 and TNFα | Baseline (day 0)
  The samples will be centrifuged and stored at -80°C. Salivary levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated by Enzyme Linked Immune Sorbent Assay (ELISA), according to manufacturer's instructions.
Salivary levels of IL-1β, IL-6, IL-8, IL-10 and TNFα | After 4 weeks of treatment (Day 30)
  The samples will be centrifuged and stored at -80°C. Salivary levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated by Enzyme Linked Immune Sorbent Assay (ELISA), according to manufacturer's instructions.
Serum levels of IL-1β, IL-6, IL-8, IL-10 and TNFα | Baseline (Day 0)
  Peripheral blood will be centrifuged at 400xg for 10 min at 4°C. Serum will be collected and stored at -80°C. Serum levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated by Enzyme Linked Immune Sorbent Assay (ELISA), according to manufacturer's instructions.
Serum levels of IL-1β, IL-6, IL-8, IL-10 and TNFα | After 4 weeks of treatment (Day 30)
  Peripheral blood will be centrifuged at 400xg for 10 min at 4°C. Serum will be collected and stored at -80°C. Serum levels of IL-6, IL-10, IL-1β, INF-γ and TNF-α will be evaluated by Enzyme Linked Immune Sorbent Assay (ELISA), according to manufacturer's instructions.
Assessment of Quality of life in OLP patients | Baseline (Day 0)
  Patient quality of life will be measured by means of the Oral Health Impact Profile (OHIP 14)
Assessment of Quality of life in OLP patients | After 4 weeks of treatment (Day 30)
  Patient quality of life will be measured by means of the Oral Health Impact Profile (OHIP 14)
Assessment of Quality of life in OLP patients | 30 days after the discontinuation of treatment (follow-up period)
  Patient quality of life will be measured by means of the Oral Health Impact Profile (OHIP 14)
Assessment of Quality of lifein OLP patients | 60 days after the discontinuation of treatment (follow-up period)
  Patient quality of life will be measured by means of the Oral Health Impact Profile (OHIP 14)
Anxiety and Depression | Baseline (Day 0)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | Participants will be evaluated after 1 week of treatment (Day 7)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | Participants will be evaluated after 2 weeks of treatment (Day 14)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | Participants will be evaluated after 3 weeks of treatment (Day 21)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | Participants will be evaluated after 4 weeks of treatment (Day 30)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | 30 days after the discontinuation of treatment (follow-up period)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)
Anxiety and Depression | 60 days after the discontinuation of treatment (follow-up period)
  Patient anxiety and depression will be measured by means of The Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernanda SD Rodrigues, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Scholl of Dentistry, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram Z, Abduljabbar T, Vohra F, Javed F. Efficacy of low-level laser therapy compared to steroid therapy in the treatment of oral lichen planus: A systematic review. J Oral Pathol Med. 2018 Jan;47(1):11-17. doi: 10.1111/jop.12619. Epub 2017 Aug 21. PMID 28766756
- [Background] Dillenburg CS, Martins MA, Munerato MC, Marques MM, Carrard VC, Sant'Ana Filho M, Castilho RM, Martins MD. Efficacy of laser phototherapy in comparison to topical clobetasol for the treatment of oral lichen planus: a randomized controlled trial. J Biomed Opt. 2014 Jun;19(6):068002. doi: 10.1117/1.JBO.19.6.068002. PMID 24887747
- [Background] Sulewska M, Duraj E, Sobaniec S, Graczyk A, Milewski R, Wroblewska M, Pietruski J, Pietruska M. A clinical evaluation of the efficacy of photodynamic therapy in the treatment of erosive oral lichen planus: A case series. Photodiagnosis Photodyn Ther. 2017 Jun;18:12-19. doi: 10.1016/j.pdpdt.2017.01.178. Epub 2017 Jan 22. PMID 28119140
- [Background] DeLand MM, Weiss RA, McDaniel DH, Geronemus RG. Treatment of radiation-induced dermatitis with light-emitting diode (LED) photomodulation. Lasers Surg Med. 2007 Feb;39(2):164-8. doi: 10.1002/lsm.20455. PMID 17311276
- [Background] Nogueira PA, Carneiro S, Ramos-e-Silva M. Oral lichen planus: an update on its pathogenesis. Int J Dermatol. 2015 Sep;54(9):1005-10. doi: 10.1111/ijd.12918. Epub 2015 Jul 3. PMID 26147778
- [Background] Alrashdan MS, Cirillo N, McCullough M. Oral lichen planus: a literature review and update. Arch Dermatol Res. 2016 Oct;308(8):539-51. doi: 10.1007/s00403-016-1667-2. Epub 2016 Jun 27. PMID 27349424
- [Background] Thongprasom K, Luangjarmekorn L, Sererat T, Taweesap W. Relative efficacy of fluocinolone acetonide compared with triamcinolone acetonide in treatment of oral lichen planus. J Oral Pathol Med. 1992 Nov;21(10):456-8. doi: 10.1111/j.1600-0714.1992.tb00974.x. PMID 1460584
- [Background] Lilleby K, Garcia P, Gooley T, McDonnnell P, Taber R, Holmberg L, Maloney DG, Press OW, Bensinger W. A prospective, randomized study of cryotherapy during administration of high-dose melphalan to decrease the severity and duration of oral mucositis in patients with multiple myeloma undergoing autologous peripheral blood stem cell transplantation. Bone Marrow Transplant. 2006 Jun;37(11):1031-5. doi: 10.1038/sj.bmt.1705384. PMID 16633359
- [Background] Carrozzo M, Gandolfo S, Lodi G, Carbone M, Garzino-Demo P, Carbonero C, Porter SR, Scully C. Oral lichen planus in patients infected or noninfected with hepatitis C virus: the role of autoimmunity. J Oral Pathol Med. 1999 Jan;28(1):16-9. doi: 10.1111/j.1600-0714.1999.tb01988.x. PMID 9890452
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Derived] Sobral SS, da Silva Brandao EH, de Barros Gallo C, Molon A, Sobral APT, de Fatima Teixeira da Silva D, Motta LJ, Dos Santos Franco AL, Rodrigues MFSD. Analysis of the psychopathological profile, quality of life, and cost-effectiveness of oral lichen planus patients treated with photobiomodulation. Clin Oral Investig. 2022 Jan;26(1):719-728. doi: 10.1007/s00784-021-04050-z. Epub 2021 Jul 12. PMID 34251533
- [Derived] Ferri EP, Gallo CB, Abboud CS, Yanaguizawa WH, Horliana ACRT, Silva DFTD, Pavani C, Bussadori SK, Nunes FD, Mesquita-Ferrari RA, Fernandes KPS, Rodrigues MFSD. Efficacy of photobiomodulation on oral lichen planus: a protocol study for a double-blind, randomised controlled clinical trial. BMJ Open. 2018 Oct 8;8(10):e024083. doi: 10.1136/bmjopen-2018-024083. PMID 30297352